CLINICAL TRIAL: NCT00206817
Title: Rapid Assessment of Cardiac Markers for the Evaluation of Acute Coronary Syndrome (RACE-ACS)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott RDx Cardiometabolic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 020
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

INTERVENTIONS:
Device: Triage CardioProfilER (Troponin I, Myoglobin, CK-MB, BNP)

SUMMARY:
This clinical trial is being conducted to 1) evaluate the possible usefulness of a panel of cardiac markers in assessing emergency department patients with possible acute coronary syndrome, 2) evaluate the usefulness of BNP in assessing emergency department patients with possible acute coronary syndrome, 3) determine if BNP can be used to predict adverse events during hospitalization and in the emergency department, and 4) evaluate how a Point-of-Care testing platform affects resource utilization in the emergency department.

DETAILED DESCRIPTION:
The correct diagnosis of acute coronary syndrome (ACS) remains a frequent significant challenge for emergency physicians. Over eight million chest pain patients present annually and despite promising advances in diagnosis, over four percent of ACS patients are mistakenly discharged home. While the history and physical, cardiac risk factor assessment, ECG, and cardiac marker determination are all included in the assessment and risk stratification of patients presenting with possible ACS, this assessment is clearly far from perfect. Improved rapid and accurate means of assessment in this population in the ED are clearly needed.ED patients with chest discomfort will be screened and approached for study enrollment. Consenting patients meeting the study inclusion and exclusion criteria will be enrolled. Point-of-care serial cardiac marker measurements will be performed. Based on a web-based computerized randomization system, half (50%) the patients willundergo routine central laboratory testing only. Half (50%) of the patients will undergopoint-of-care markers performed in the ED in addition to routine central laboratory testing.In this second group, central laboratory test results will be blinded from the ED physicianuntil the disposition time. BNP will be blinded and not reported to physicians for the first 500 patients (Phase I). After the first 500 patients have been enrolled, an interim analysis will be performed to determine the clinical utility of BNP in patient assessment. After physician education of these results, the trial will resume for the remaining 500 patients (Phase II). In Phase II, BNP levels will be provided to the physicians using the same time and randomization format.The patients and their medical records will be followed for a period of thirty days and sixmonths after enrollment.

ELIGIBILITY:
Inclusion Criteria:

Age greater than or equal to 21 years at the time of enrollment Chest discomfort or other symptoms consistent with possible ACS as indicated by the treating physician obtaining an ECG and cardiac markers for the patient's evaluation New onset or worsening symptoms within six hours of presentation to the ED.

Exclusion Criteria:

History of CHF per patient history or in the available medical record. History of end stage renal disease on dialysis. Refused informed consent.4) Refused medical record review and telephone follow up at 30 days and six months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-10

PRIMARY OUTCOMES:
Sensitivity and specificity of the three-marker versus the four-marker panelDetermine the added benefit of BNP in the diagnosis of patients with ACS

SECONDARY OUTCOMES:
Determine the economic and resource utilization benefit of the POC platform vs. standard lab testing

CONTACTS AND LOCATIONS:
Overall Officials: Andra L Blomkalns, MD, Principal Investigator — University of Cinncinati
Locations (6):
- United States (6):
  - UC Davis Medical Center, Sacramento, California
  - Henry Ford Health Systems, Detroit, Michigan
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Univ. Baptist Med. Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation Dept. of Emergency Medicine, Cleveland, Ohio